CLINICAL TRIAL: NCT01602211
Title: INSPIRE for Survivorship After Transplant: A Multicenter Randomized Controlled Trial of an Internet and Social-Media Program for Long-Term Hematopoietic Cell Transplantation Survivors
Brief Title: INSPIRE: Internet and Social-media Program With Information and Resources for Long-Term Cancer Survivors Who Underwent Stem Cell Transplant
Acronym: INSPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2605.00; NCI-2012-00743 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2605.00 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA160684 (NIH)
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2017-09

CONDITIONS: Cancer Survivor; Depression; Hematopoietic and Lymphoid Cell Neoplasm; Myelodysplastic Syndrome
Keywords: stem cell transplant; cancer survivors; internet; social media; distress; health care adherence
MeSH Terms: conditions — Depression; Hematologic Neoplasms; Myelodysplastic Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (INSPIRE internet full program access) (Experimental): Participants receive full access to the INSPIRE internet site comprising an individually tailored program with a greeting home page with links to each target area, a 'My Health Action Plan' health care guideline for transplant survivors, self-care tips and tool pages for each complication and major issues for HCT survivors, a section for each complication (mood, energy, heart health, strengthening bones, second cancers), resource pages, opportunities to send secure messages with questions or comments on any topic, opportunities to request additional assistance or information, mobile texting options, and social media links (Twitter/Facebook/Pinterest) maintained and monitored by the Social Media Specialist.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (delayed program access control) (Experimental): Participants receive annotated website links to existing transplant and cancer survivor sites, followed by delayed access to the INSPIRE internet program after 1 year.
  Interventions: Other: Internet-Based Intervention; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Receive full access to INSPIRE
  Arms: Arm I (INSPIRE internet full program access)
Other: Internet-Based Intervention — Receive access to an annotated list of existing resources for transplant and cancer survivors and delayed access to INSPIRE site
  Arms: Arm II (delayed program access control)
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
  Arms: Arm II (delayed program access control)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies an internet and social-media program for improving quality of life in long-term survivors who underwent stem cell transplant. In this study, researchers want to compare a survivorship internet program to the standard treatment of currently available internet sites for transplant survivors to learn which works better for people who have received bone marrow or blood stem cell transplants. A survivorship-focused internet program may improve mood, stress, and preventive health care, and provide useful health resources for transplant survivors. It is not yet known whether currently available internet sites are more effective than a survivorship-focused internet program in improving quality of life in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether 2-10 year hematopoietic cell transplant (HCT) survivors with elevated depression or cancer-related distress who are randomized to receive access to a tailored internet-based program report reduced depression and distress when compared with control group survivors who receive access to an internet site with links to transplant and cancer-specific online resources and delayed access to the internet site (active control).

II. Determine whether survivors with low survivorship preventive care adherence (PCA) who are randomized to receive access to the tailored internet-based program, including a survivorship preventive care plan, report increased PCA when compared with the active control group survivors.

SECONDARY OBJECTIVES:

I. Secondary outcomes will include process measures of internet study reach and utilization, as well as physical function, physical activity level, and knowledge of survivorship needs. Further analyses will identify risk factors for disparities in survivorship preventive care adherence in HCT survivors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Participants receive full access to the INSPIRE internet site comprising an individually tailored program with a greeting home page with links to each target area, a 'My Health Action Plan' health care guideline for transplant survivors, self-care tips and tool pages for each complication and major issues for HCT survivors, a section for each complication (mood, energy, heart health, strengthening bones, second cancers), resource pages, opportunities to send secure messages with questions or comments on any topic, opportunities to request additional assistance or information, mobile texting options, and social media links (Twitter/Facebook/Pinterest) maintained and monitored by the Social Media Specialist.

ARM II: Participants receive annotated website links to existing transplant and cancer survivor sites, followed by delayed access to the INSPIRE internet program after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Received a transplant at a consortium center for a hematologic malignancy or myelodysplasia
* Currently 2-10 years after first HCT

Exclusion Criteria:

* Does not have internet and email access; note that survivors otherwise eligible, but excluded from full study participation because of this exclusion, will be asked to fill out a mailed copy of the baseline assessment for use in secondary aims analyses; they will be sent an information form and a copy of the tailored 'My Health Action Plan' health care guideline for transplant survivors also provided to randomized participants
* English insufficient to complete baseline patient-reported outcomes (PRO) assessments
* Has received treatment for a recurrent or 2nd cancer that required > surgical excision in the past 2 years or did not have a hematologic malignancy or myelodysplasia diagnosis or did not receive a first transplant between 2-10 years before approach for the study; (these participants will be ineligible for randomization, but will have intervention site access if they complete baseline PRO assessment)
* Scores 20 or above on the patient health questionnaire (PHQ)-8 depression measure (indicating severe depression); these participants will be contacted by a study psychologist to evaluate and provide resources to address their needs (2% of enrollees in our previous study); they will be ineligible for randomization, but will have intervention site access if they complete baseline PRO assessment
* Residing in an institution or other living situation where health care decisions are not made by the participant (e.g., hospitalized, prisoners, living in a rehabilitation facility)
* Does not complete baseline PRO assessment items required to determine stratification or whether the survivor meets inclusion and exclusion criteria
* Has medical or health issues prohibiting computer use (e.g., vision-impaired, cognitively impaired, illness or accident impairing computer function)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2013-05-14 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Cancer and treatment distress (CTXD) score as reported on the PCA using binary outcomes | Up to 12 months
PHQ-8 depression score as reported on the PCA, using binary outcomes | Up to 12 months
Proportion of adherence to recommended survivorship preventive care and barriers to PCA | Up to 12 months

SECONDARY OUTCOMES:
Health behaviors | Up to 12 months
  Composite measure of health behaviors, including tobacco use, alcohol use, physical activity, use of sunscreen, food intake, body mass index, and sleep.
Physical function, as assessed by the Patient Reported Outcomes Measurement Information System scale | Up to 12 months
Total minutes per week of moderate to vigorous intensity exercise as assessed by the Godin Leisure Time Exercise Questionnaire | Up to 12 months
  This measure is a measure of leisure time physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Syrjala, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Farhadfar N, Weaver MT, Al-Mansour Z, Yi JC, Jim HSL, Loren AW, Majhail NS, Whalen V, Uberti J, Wingard JR, Lynch Kelly D, Syrjala KL. Self-Efficacy for Symptom Management in Long-Term Adult Hematopoietic Stem Cell Survivors. Transplant Cell Ther. 2022 Sep;28(9):606.e1-606.e8. doi: 10.1016/j.jtct.2022.05.035. Epub 2022 May 31. PMID 35662590
- [Derived] Banerjee R, Yi JC, Majhail NS, Jim HSL, Uberti J, Whalen V, Loren AW, Syrjala KL. Driving Distance and Patient-Reported Outcomes in Hematopoietic Cell Transplantation Survivors. Biol Blood Marrow Transplant. 2020 Nov;26(11):2132-2138. doi: 10.1016/j.bbmt.2020.08.002. Epub 2020 Aug 8. PMID 32781287